CLINICAL TRIAL: NCT04561336
Title: CAVE (Cetuximab-AVElumab) mCRC: A Single Arm Phase II Clinical Study of the Combination of Avelumab Plus Cetuximab in Pre-treated RAS Wild Type Metastatic Colorectal Cancer Patients
Brief Title: Avelumab Plus Cetuximab in Pre-treated RAS Wild Type Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Fortunato Ciardiello, Full Professor, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS 100070-0028; 2017-004392-32 (EudraCT Number)
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Colorectal Cancer; RAS Wild Type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — avelumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: combination treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- avelumab plus cetuximab (Experimental): avelumab at a dose of 10 mg/kg once every 2 weeks plus cetuximab at a starting dose of 400 mg/m2 by i.v.infusion over 120 minutes at first dose and at the dose of 250 mg/ m2 by i.v.infusion over 60 minutes for subsequent infusions every week.
  Interventions: Drug: Avelumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Avelumab — avelumab in combination with cetuximab
Drug: Cetuximab — avelumab in combination with cetuximab

SUMMARY:
This is a non-profit phase II, open-label, single-arm study of cetuximab plus avelumab in patients with RAS WT mCRC treated in first line with chemotherapy in combination with an anti- EGFR drug that have had a clinical benefit (complete or partial response) from treatment.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy (OS) of avelumab and cetuximab combined in pre-treated RAS wild type metastatic colorectal cancer patients. Tumor measurements by computed tomography (CT) scan or magnetic resonance imaging (MRI) will be performed every 8 weeks from the beginning of treatment to determine response to treatment. Response will be evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

Treatment will continue until disease progression, significant clinical deterioration, unacceptable toxicity, any criterion for withdrawal from the trial or trial drug is fulfilled. Treatment may continue past the initial determination of disease progression per RECIST 1.1 if the subject's performance status has remained stable, and if in the opinion of the Investigator, the subject will benefit from continued treatment and if other criteria are fulfilled as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before any trial-related procedure is undertaken that is not part of the standard patient management
2. Male or female subjects aged ≥ 18 years 3.Histologically proven diagnosis of colorectal adenocarcinoma.

4. Diagnosis of metastatic disease 5. RAS (NRAS and KRAS exon 2,3 and 4) wild-type in tissue at initial diagnosis. 6. Efficacy of a first line therapy containing an anti-EGFR agent (panitumumab or cetuximab) with a major response achieved (complete or partial response).

7. A second line therapy. 8. More than 4 months from last dose of anti-EGFR agent administered in first line treatment before randomization. 9.Measurable disease according to RECIST criteria v1.1 10 ECOG PS of 0 to 1 at trial entry 11. Estimated life expectancy of more than 12 weeks 12. Adequate hematological function defined by white blood cell (WBC) count ≥ 2.5 × 109/L with absolute neutrophil count (ANC) ≥ 1.5 × 109/L, lymphocyte count ≥ 0.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused) 13. Adequate hepatic function defined by a total bilirubin level

≤ 1.5 × the upper limit of normal (ULN) range and AST and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN for all subjects or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).

14. Adequate renal function defined by an estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) 15. Effective contraception for both male and female subjects if the risk of conception exists (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use effective contraception, defined as 2 barrier methods, or 1 barrier method with a spermicide, an intrauterine device, or use of oral female contraceptive. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately.) Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists.

16. No prior immunotherapy

Exclusion Criteria:

Subjects are not eligible for this trial if they fulfill any of the following exclusion criteria:

1. Any contraindication to cetuximab and/or avelumab.
2. Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix.
3. Pregnancy 4.Breastfeeding

5. Participation in a clinical study or experimental drug treatment within 30 days.

6. Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the trial treatment, with the exception of:

* subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to

  ≤ 10 mg prednisone daily
* intranasal, inhaled, topical steroids,
* local steroid injection (e.g., intra-articular injection)
* Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) 7. All subjects with brain metastases, except those meeting the following criteria:
* Brain metastases have been treated locally, and
* No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable) 8. Prior organ transplantation, including allogeneic stem-cell transplantation 9. Significant acute or chronic infections including, among others:
* Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive) 10. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:
* Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
* Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or equivalent prednisone per day.
* Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable.
* Active infection requiring systemic therapy. 11. Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon is acceptable as long as it is anticipated that the administration of steroids will be completed in 14 days, or that the daily dose after 14 days will be ≤ 10 mg per day of equivalent prednisone.

  12. Known severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more feauters of partially controlled asthma).

  13. History of hypersensitivity to Polysorbate 80 that led to unacceptable toxicity requiring treatment cessation 14. Persisting toxicity related to prior therapy of Grade > 1 NCI- CTCAE v 4.03.

  15. Known alcohol or drug abuse. 16. Clinically significant (that is active) cardioavscular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, comgestive heart failure (New York Heart Association Classification Class≥II), or serious uncontrolled cardiac arrhytmia requiring medication 17. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

  18. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.

  19.Vaccination within 4 weeks of the first dose of avelumab and cetuximab and while on treatment is prohibited except for administration of inactivated vaccine (i.e. inactivated influenza vaccine) 20. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Ciardiello, MD, Principal Investigator — Università della Campania L Vanvitelli
Locations (1):
- Università della Campania Luigi Vanvitelli, Napoli, Italy

REFERENCES:
- [Derived] Ciardiello D, Martinelli E, Troiani T, Mauri G, Rossini D, Martini G, Napolitano S, Famiglietti V, Del Tufo S, Masi G, Santini D, Avallone A, Pietrantonio F, Lonardi S, Di Maio M, Zampino MG, Fazio N, Bardelli A, Siena S, Cremolini C, Sartore-Bianchi A, Ciardiello F. Anti-EGFR Rechallenge in Patients With Refractory ctDNA RAS/BRAF wt Metastatic Colorectal Cancer: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245635. doi: 10.1001/jamanetworkopen.2024.5635. PMID 38592721
- [Derived] Martini G, Ciardiello D, Famiglietti V, Rossini D, Antoniotti C, Troiani T, Napolitano S, Esposito L, Latiano TP, Maiello E, Del Re M, Lonardi S, Aprile G, Santini D, Masi G, Avallone A, Normanno N, Pietrantonio F, Pinto C, Ciardiello F, Cremolini C, Martinelli E. Cetuximab as third-line rechallenge plus either irinotecan or avelumab is an effective treatment in metastatic colorectal cancer patients with baseline plasma RAS/BRAF wild-type circulating tumor DNA: Individual patient data pooled analysis of CRICKET and CAVE trials. Cancer Med. 2023 Apr;12(8):9392-9400. doi: 10.1002/cam4.5699. Epub 2023 Mar 7. PMID 36880426
- [Derived] Martinelli E, Martini G, Famiglietti V, Troiani T, Napolitano S, Pietrantonio F, Ciardiello D, Terminiello M, Borrelli C, Vitiello PP, De Braud F, Morano F, Avallone A, Normanno N, Nappi A, Maiello E, Latiano T, Falcone A, Cremolini C, Rossini D, Santabarbara G, Pinto C, Santini D, Cardone C, Zanaletti N, Di Liello A, Renato D, Esposito L, Marrone F, Ciardiello F. Cetuximab Rechallenge Plus Avelumab in Pretreated Patients With RAS Wild-type Metastatic Colorectal Cancer: The Phase 2 Single-Arm Clinical CAVE Trial. JAMA Oncol. 2021 Oct 1;7(10):1529-1535. doi: 10.1001/jamaoncol.2021.2915. PMID 34382998